CLINICAL TRIAL: NCT03024697
Title: Single-shot Pectoral Plane (PECs) Blocks Versus Continuous Local Anaesthetic Infusion Analgesia or Both PECs Block and Local Anaesthetic Infusion After Non-ambulatory Breast Cancer Surgery: A Prospective, Randomised, Double-blind Trial
Brief Title: Single-shot Pectoral Plane(PECs) Block Versus Continuous Local Anaesthetic Infusion Analgesia or Both PECS Block and Local Anaesthetic Infusion After Breast Surgery: A Prospective Randomised, Double-blind Trial
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mater Misericordiae University Hospital (Other)
Responsible Party: Principal Investigator, Sean Keane, Dr. Sean Keane; Anaesthesia SpR, Mater Misericordiae University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: PECS 123
Record Dates: First submitted 2017-01-15; First posted 2017-01-19 (Estimated); Last update posted 2017-09-11 (Actual); Status verified 2017-09

CONDITIONS: Breast Diseases; Anesthesia; Block
Keywords: Breast surgery; Pectoral plane block; PECs; Local anaesthesia infusion; Analgesia
MeSH Terms: conditions — Breast Diseases; Bites and Stings; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PECs Block (Active Comparator): Patients randomised to receive pectoral plane blocks and a sham local anaesthetic infusion wound catheter
  Interventions: Procedure: Pectoral Plane Block
- LA Infusion (Active Comparator): Patients randomised to receive a local anaesthetic infusion wound catheter; No sham pectoral plane block performed as patients usually under general anaesthetic at time of block.
  Interventions: Procedure: Local Anaesthetic Wound Infusion Catheter
- PECs Block & LA Infusion (Active Comparator): Patients randomised to receive pectoral plane blocks and a local anaesthetic infusion wound catheter.
  Interventions: Procedure: Pectoral Plane Block; Procedure: Local Anaesthetic Wound Infusion Catheter

INTERVENTIONS:
Procedure: Pectoral Plane Block
  Other Names: PECs Block
  Arms: PECs Block; PECs Block & LA Infusion
Procedure: Local Anaesthetic Wound Infusion Catheter — Levobupivicaine 0.1% @10ml/hr via a wound infusion catheter
  Other Names: Local Anaesthetic Infusion
  Arms: LA Infusion; PECs Block & LA Infusion

SUMMARY:
In this proposed study, the investigators are looking to conduct a prospective, randomised, double-blind, non-inferiority trial, to study single-shot pectoral plane (PECs) blocks versus continuous local anaesthetic infusion analgesia versus a combination of PECs blocks and local anaesthetic infusion analgesia, when it comes to providing analgesia for most forms of breast surgery.

Breast surgery is common, and the optimal form of analgesia is currently unknown. Techniques involving local anaesthetic, such as pectoral plane (PECs) blocks and infusion pumps, are growing in popularity, as they reduce the amount of opioid medications used. Opioids are associated with nausea, vomiting, low blood pressure, drowsiness and constipation, and as such, opioid-sparing analgesic regimens postoperatively are becoming more common. These regimens will typically involve paracetamol, a NSAID (non-steroidal anti-inflammatory drug), and a local anaesthetic technique.

Pectoral plane blocks involve a once-off injection of local anaesthetic at two locations within the chest wall, typically done after the patient undergoes general anaesthesia, but before the commencement of surgery. Local anaesthetic infusion pumps involve the insertion of a catheter into the wound at the end of surgery, before the patient emerges from general anaesthesia, that constantly emit local anaesthetic over a defined period of time. Each technique is considered extremely safe, and is considered acceptable as a form of pain relief in patients undergoing breast surgery.

There are no published works comparing pectoral plane blocks with local anaesthetic infusion pump analgesia, and the investigators see a gap in the knowledge base that can be addressed. This study will allow efficacy, safety and cost of the three techniques to be compared. The investigators feel the study design is robust, and statistical analysis based on previously published works in the area of postoperative analgesia has allowed the study to be powered appropriately.

Patients undergoing breast surgery are a vulnerable group, and this is recognised via the provision of a comprehensive Patient Information Leaflet and a commitment to respecting the process of Informed Consent. The investigators also recognise this is a stressful period in a woman's life, and the study will be conducted in a sensitive and compassionate manner.

The study has been designed to be prospective, randomised, and double-blinded. The anaesthetic will be standardised in relation to analgesic and anti-emetic agents administered, in order to minimise variables. Chronic post-surgical pain is a growing area of research, and the follow-up telephone interview at 3-months will allow investigation of this.

A Data Record Form will be utilised for data collection, which will subsequently be analysed statistically. Data will be handled sensitively, securely, and by the minimum number of researchers. A plan is in place for destruction of data at an appropriate time.

While there will be no direct benefit to participants, including monetary considerations, this research study will add to the knowledge-base surrounding analgesia for breast surgery.

DETAILED DESCRIPTION:
Methods The Mater Misericordiae University Hospital's Institutional Review Board (IRB) approved this study; reference number 1/378/1840, dated December 21st, 2016. It was registered with clinicaltrials.gov; reference number NCT03024697, dated February 15th, 2017. Forty-five ASA I-III female patients aged 18 years or older, undergoing non-ambulatory breast cancer surgery under general anaesthesia between January and May 2017 were included. All participants provided informed written consent.

Non-ambulatory breast cancer surgery encompassed wide-local excision with lymph node resection, simple mastectomy, and mastectomy with lymph node resection. Those undergoing latissimus dorsi or DIEP (deep inferior epigastric perforator) flap reconstruction were excluded. Patients with chronic pain syndromes, local anaesthetic allergy, contraindication to simple analgesics, local infection over the proposed block site, coagulopathy, or co-morbid conditions precluding the provision of informed consent, were excluded. All patients were day of surgery admission and attended a preoperative anaesthetic assessment clinic.

Patients were allocated into three groups using computer-generated randomisation, with the study number and group allocation concealed in sealed envelopes. Blocked randomisation in groups of 9 was applied, giving similar numbers in each group as the study progressed. Groups were named 'PECs', 'Local anaesthetic infusion (LA infusion)' , and 'Both (PECS & LA infusion)', which were evenly distributed to opaque envelopes numbered one to forty-five in accordance with randomisation. The randomisation key was held by an independent party, and was not used to reveal participant group allocations until data analysis commenced. 'PECs' patients received PECS I & II blocks and a sham wound infiltration catheter. 'LA infusion' patients received a continuous local anaesthetic wound infusion catheter. 'PECs & LA infusion' patients received a combination of techniques, without the initial local anaesthetic bolus via the wound infusion catheter. PECs blocks were performed while patients were under general anaesthesia, prior to the commencement of surgery. The operative surgeon sited wound infusion catheters during skin closure at the end of surgery.

Patients were induced with fentanyl 1-2 μg.kg-1, followed by propofol titrated to the absence of verbal response. Anaesthesia was maintained using an oxygen, air and sevoflurane combination. Airway management and lung ventilation strategies were at the discretion of the supervising anaesthetist. Patients received a standard intraoperative analgesic regimen of paracetamol 1g and dexketoprofen 50mg intravenously (IV), with rescue morphine as deemed necessary. Combination antiemetics, including ondansetron 0.1-0.15 mg.kg-1 IV, dexamethasone 0.1-0.2 mg.kg-1 IV or droperidol 0.01-0.015 mg.kg-1 IV, were administered according to patient risk factors. Intraoperative management was otherwise left to the discretion of the supervising anaesthetist. Routine monitoring was used in accordance with AAGBI guidelines15. An electronic anaesthetic record was used to document physiological parameters. Perioperative events, such as induction of anaesthesia, initial skin incision, and end of surgery, were annotated on the record.

PECs I & II blocks were performed on the side of surgery, using the ultrasound-guided technique described by Blanco et al9, 10. The patient was placed in the supine, head-up, position with the arm abducted. The skin was prepared with chlorhexidine gluconate 2%/isopropyl alcohol 70% (BD, ChloraPrep, NJ, USA). PECs blocks were performed with a 22-gauge echogenic needle (B. Braun, Ultraplex 360 cannula, Hessen, Germany; 50-80mm), using the same ultrasound machine (Sonosite Edge, Sonosite, Inc., Bothwell, WA, USA) and transducer (Sonosite HFL 50x, Sonosite, Inc., Bothwell, WA, USA). The ultrasound probe was placed inferolaterally at the mid-clavicular level. The axillary artery and vein were identified, and the probe moved laterally until pectoralis major, pectoralis minor and serratus anterior muscles were located at the level of the 3rd rib. A needle in-plane approach was taken until the needle tip was positioned in the plane between pectoralis major and minor muscles, and levobupivacaine 0.25% 10ml was injected. The needle was advanced until it occupied the space between pectoralis minor and serratus anterior muscles, and a further 20ml of levobupivacaine 0.25% was injected.

Blinding was not considered necessary for 'LA infusion' group patients, as PECs blocks were performed under general anaesthesia. All patients had a wound infusion catheter sited and attached to an elastometric pump (B. Braun, ON-Q PainBuster, Hessen, Germany), which was placed by the operating surgeon during skin closure at the end of surgery. For blinding purposes, patients in the 'PECs' group received a sham wound infiltration catheter system. 'LA infusion' and 'PECS & LA infusion' patients received levobupivacaine 0.1% at 10ml.hr-1 for 24 hours postoperatively, while 'PECs' patients received sodium chloride 0.9% at the same rate. 'LA infusion' patients were administered an initial bolus of levobupivacaine 0.25% 20ml at the end of surgery. Those who performed the procedures, or were involved in the perioperative management, were not involved in postoperative pain assessment or data collection. Study interventions as described occurred while patients were under general anaesthesia.

Patients were monitored for 24 hours after surgery, initially in the post-anaesthesia care unit (PACU), and then at ward level once PACU discharge criteria were met. Oxycodone 1-2mg IV as required was prescribed for rescue analgesia in the PACU. A standard analgesic protocol of paracetamol 1g PO/IV 6-hourly regular, ibuprofen 400mg PO 8-hourly regular, and oxycodone immediate release (oxynorm) 5-10mg 1-hourly as required for rescue analgesia, was prescribed for all patients. Ondansetron 4-8mg IV 8-hourly as required was prescribed, to be administered in the event of postoperative nausea and vomiting (PONV).

The primary outcome measure of the study was area under curve of verbal rating score (VRS) of pain moving versus time, (AUC) where VRS pain was measured at 1 hour, 4-6 hours, 10-14 hours, and 20-24 hours postoperatively. At each assessment, patients were invited to report their pain VRS pain at rest. Pain while moving was defined as pain experienced while sitting forward from a recumbent position. Secondary outcome measures were total opioid consumption over a 24-hour period and presence of adverse events. An investigator masked to group allocations recorded vital signs, pain scores, antiemetic administration and opioid use postoperatively. Adverse events such as sedation, respiratory depression, hypotension, pruritus and PONV were also recorded.

Statistical Analysis

Data was analysed by Graph Pad Prism v6 (Salt Lake City, UH). The primary end-point was area under the VRS moving versus time curve (AUC). We powered the study to detect a 25% difference in AUC from an internal pilot study which indicated mean AUC of 60 cm.hr-1 (SD 5-10) among patients receiving PECs or LA infusion in our clinical service, to 45 cm.hr-1. We had observed the standard deviation of the AUC to be in the order of 15 cm.hr-1. Assuming a Type I error of 0.05 and a Type II error of 0.1, then n=11 patients would be required each group to detect this difference with 90% power. We obtained IRB permission for n=15 each group to allow for protocol violations or patient drop-out.

Data was collected at 1, 4-6, 12-14 and 20-24 hr, post-operatively. It was tested for distribution initially using the Kolmogorov-Smirnov test. For each patient, their AUC both moving and at rest was calculated by plotting their pain VRS versus time using Graph Pad Prism v.6. The mean AUC according to the three study groups was then calculated and inspected for distribution as described above, and all AUC data was found to be normally distributed. Therefore, AUC data is expressed as mean ± SD and was compared using ANOVA with post hoc Bonferroni correction. Non-normally distributed data was compared using the Kruskal-Wallis test for repeated measurements. Categorical data (e.g. the incidence of potential adverse effects) were compared using Fischer's exact test where appropriate. P<0.05 was deemed statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Undergoing breast surgery, including wide local excision (WLE) and sentinel lymph node biopsy (SLNB), mastectomy +- SLNB

Exclusion Criteria:

* Male
* Undergoing flap reconstruction breast surgery, implant surgery or bilateral breast surgery
* Chronic pain syndrome
* Local anaesthetic allergy
* Contraindication to routine postoperative analgesia, e.g. paracetamol
* Contraindication to regional anaesthesia, i.e. localised infection

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Area under curve of verbal rating score (VRS) of pain moving versus time | VRS pain was measured at 1 hour, 4-6 hours, 10-14 hours, and 20-24 hours postoperatively

SECONDARY OUTCOMES:
Total postoperative opioid consumption | Over first 24 postoperative hours
Postoperative nausea and vomiting | Recorded at the following time points after surgery: 1 hour, 2-4 hours, 6-8 hours, 10-14 hours 20-24 hours
Postoperative sedation score | Recorded at the following time points after surgery: 1 hour, 2-4 hours, 6-8 hours, 10-14 hours 20-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Donal Buggy, Principal Investigator — Mater Misericordiae University Hospital
Locations (1):
- Department of Anaesthesia, Mater Misericordiae University Hospital, Dublin, Ireland

IPD SHARING:
Plan to Share IPD: No
IPD will not be made available to other researchers as this has been pre-determined with patients as part of the process of informed consent.

REFERENCES:
- [Derived] O'Scanaill P, Keane S, Wall V, Flood G, Buggy DJ. Single-shot pectoral plane (PECs I and PECs II) blocks versus continuous local anaesthetic infusion analgesia or both after non-ambulatory breast-cancer surgery: a prospective, randomised, double-blind trial. Br J Anaesth. 2018 Apr;120(4):846-853. doi: 10.1016/j.bja.2017.11.112. Epub 2018 Feb 14. PMID 29576125